CLINICAL TRIAL: NCT04065503
Title: Detection and Persistence of a Product Containing L. Helveticus R-0052, L. Casei HA-108, B. Breve HA-129, B. Longum R-0175 and S. Thermophilus HA-110 in Healthy Adults: an Open-label Pilot Study.
Brief Title: Probiotic Detection and Persistence Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Lallemand Health Solutions, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB201902202; OCR26142 (Other: UF OnCore); AGR00015606 (Other: UFIRST)
Record Dates: First submitted 2019-08-20; First posted 2019-08-22 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Healthy
Keywords: probiotic; gut transit time

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Adults (Experimental): Healthy adults will be given probiotic strains to evaluate the detection and persistence of the strains in the participant's feces.
  Interventions: Biological: Probiotic Strains

INTERVENTIONS:
Biological: Probiotic Strains — A commercial product containing L. helveticus R0052, L. casei HA-108, B. breve HA-129, and B. longum R0175 and S. thermophilus HA-110 be given to healthy adults across a 10-week open label pilot study.

SUMMARY:
The aims of this study are to determine how long it takes for the strains of a probiotic formulation to be detected in feces after the start of an intervention, how long they persist after the end of the intervention, and the associations between detection and persistence with total gut transit time.

DETAILED DESCRIPTION:
This is a 10-week interventional, open-label pilot study designed to evaluate the detection and persistence of L. helveticus R-0052, L. casei NI319, B. breve NI337, and B. longum R-0175 strains in feces of healthy adults following the start and the end of IP intervention, respectively. This study will have an initial baseline period (4 weeks), a probiotic intervention (2 weeks) and a washout period (4 weeks). Participants will complete daily questionnaires regarding stool frequency, time of stool collections, and IP intake. A weekly Gastrointestinal Symptom Rating Scale (GSRS) questionnaire will be administered. Transit time will be assessed using radiopaque markers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults ≥ 18 to < 55 years of age.
* Habitually produces at least one bowel movement per day.
* Willingness to maintain their usual diet and exercise patterns throughout the study.
* Able to provide written informed consent in English.
* Willing to provide stools and complete questionnaires, records, and diaries associated with the study and to complete all study visits.
* Willingness to discontinue consumption of probiotics and fermented products (e.g. yogurts, kombucha, fermented pickles and other fermented foods with live, active cultures) and probiotic supplements.

Exclusion Criteria:

* Elite athletes or long-distance runners.
* Concurrent consumption of fermented foods or probiotics. However, individuals will be eligible for participation after a four (4) week wash-out period.
* Known to be pregnant (self-disclosure) or breastfeeding or planning on becoming pregnant in the next 2 months.
* Use of antibiotic drugs (e.g., neomycin, rifaximin) within 1 month of the screening visit. The screened participant would be eligible to participate four (4) weeks after completing their course of antibiotics (washout period).
* Use of other investigational products within 3 months of the screening visit.
* Previously or are currently being treated for any previously or currently being treated for any intestinal disease or condition such as IBS, Crohn's disease, ulcerative colitis, celiac disease, or gastrointestinal cancer.
* Immune disorders or with possible immune deficient status (e.g. due to surgery).
* Milk or soy allergy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in time to detection of probiotic strains | Day 1; Day 2; Day 3, Day 4, Day 7, Day 10
  using strain-specific qPCR assays.
Change in time to non-detection (persistence) of probiotic strains | Day 14, Day 15, Day 16, Day 17, Day 18, Day 21, Day 24, Day 28, Day 35, Day 42
  using strain-specific qPCR assays.

SECONDARY OUTCOMES:
Whole gut transit time | Day 1, Day 2, Day 3, Day 4
  Whole gut transit time measured by radiopaque marker recovery in intervention stools

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Dahl, Principal Investigator — University of Florida
Locations (1):
- Food Science and Human Nutrition Department, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No